CLINICAL TRIAL: NCT06426160
Title: Tocilizumab for Painful Chronic Pancreatitis: A Randomised, Placebo-Controlled, Double-blinded, Investigator Initiated Trial (TOPAC Trial)
Brief Title: Tocilizumab for Painful Chronic Pancreatitis
Acronym: TOPAC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Soren Schou Olesen (Other)
Collaborators: Aarhus University Hospital (Other); University of Aarhus (Other); Viborg Regional Hospital (Other); Stanford University (Other); Haukeland University Hospital (Other)
Responsible Party: Sponsor-Investigator, Soren Schou Olesen, Professor, MD, Ph.D., Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F2024-054; 2023-510084-35-00 (EU CTIS Number)
Record Dates: First submitted 2024-05-14; First posted 2024-05-23 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Pancreatitis, Chronic
Keywords: Inflammation; Pancreatic diseases; Digestive System Diseases
MeSH Terms: conditions — Pancreatitis, Chronic; Inflammation; Pancreatic Diseases; Digestive System Diseases | interventions — tocilizumab; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomised, placebo-controlled, double-blinded investigator-initiated trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tocilizumab (Active Comparator): 8 mg / kg Tocilizumab will be diluted to a final volume of 100 mL with sterile, non-pyrogenic sodium chloride 9 mg/mL (0.9 %)
  Interventions: Drug: Tocilizumab 20 MG/ML [Actemra]
- Placebo (Placebo Comparator): 100 ml sodium chloride 9 mg/mL (0.9 %).
  Interventions: Drug: Sodium Chloride 0.9% Inj

INTERVENTIONS:
Drug: Tocilizumab 20 MG/ML [Actemra] — Tocilizumab 8 mg/kg every four weeks for 24 weeks.
  Other Names: RoActemra; Actemra
  Arms: Tocilizumab
Drug: Sodium Chloride 0.9% Inj — Placebo (Sodium chloride) every four weeks for 24 weeks.
  Other Names: Natriumchloride 0.9 % Inj
  Arms: Placebo

SUMMARY:
This placebo-controlled study will investigate the effect of tocilizumab (an anti-interleukin-6 receptor antibody) on symptom burden, physical functioning, and quality of life in patients with chronic pancreatitis.

DETAILED DESCRIPTION:
Recent independent research has emphasized the crucial role of immune cell infiltration and its interaction with pancreatic stellate cells in driving the inflammatory process and fibrogenesis in chronic pancreatitis (CP). The cytokine Interleukin 6 (IL-6) has been identified as a key mediator in this process, and preclinical studies have indicated that inhibiting IL-6 signaling can lead to favorable therapeutic outcomes. Consequently, targeting IL-6 signaling therapeutically holds great promise as a disease-modifying treatment for CP.

Until now, there have been no placebo-controlled trials in humans to test immune-modulating treatments for CP. However, there have been some promising results in preclinical studies. For example, administering an anti-IL-6 receptor antibody to an animal model of CP reduced pancreatitis-related pain, indicating a potential therapeutic effect. Blocking IL-6 signaling in an in-silico model of CP was also shown to have disease-modifying effects. Recent anecdotal evidence indicates that using tocilizumab to treat patients with COVID-19 and concomitant pancreatitis can decrease inflammation and pain in the pancreas. Additionally, blocking IL-6 signaling has been demonstrated to have anti-fibrotic effects in patients with systemic sclerosis. Taken together, these findings suggest that targeting IL-6 signaling could be a promising approach for reducing inflammation and fibrogenesis in CP. Tocilizumab (RoActemra) is an anti-IL-6 receptor antibody currently used to treat several inflammatory diseases.

Objectives:

The investigators hypothesize that treatment with tocilizumab, compared with a placebo, will reduce symptom burden (CP-related pain) and improve physical functioning and quality of life in patients with CP. In addition, the investigators hypothesize that the clinical effects will be linked to a decrease in pancreatic inflammation and fibrosis as well as systemic inflammation. The investigators also hypothesize that the pain-relieving effect of tocilizumab will lead to the normalization of pain processing in CP patients. To test these hypotheses, the project is organized into four sub-studies.

Sub-study 1 (main study - randomized placebo-controlled trial): The objective of sub-study 1 is to conduct an investigator-initiated phase 2b double-blinded, placebo-controlled, randomized clinical trial to investigate the clinical effect of tocilizumab on patient-reported outcomes.

Sub-study 2 (inflammatory biomarkers): The objective of sub-study 2 is to investigate the effects of tocilizumab on systemic inflammation using blood-based immune and fibrosis markers.

Sub-study 3 (quantitative imaging biomarkers): The objective of sub-study 3 is to investigate the effect of tocilizumab on pancreatic inflammation and fibrosis using Magnetic Resonance Imaging (MRI) of the pancreas.

Sub-study 4 (pain processing): The objective of sub-study 4 is to investigate the effect of tocilizumab on pain processing using Pancreatic Quantitative Sensory Testing (P-QST) and electrophysiological methods (EEG and ECG).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Probable or definitive diagnosis of CP according to the M-ANNHEIM criteria. This entails a typical clinical history of CP, including recurrent pancreatitis or abdominal pain in combination with the following additional criteria:
* A definitive diagnosis of CP is established by one or more of the following additional criteria:
* i) Pancreatic calcification
* ii) Moderate or marked ductal lesions (according to the Cambridge classification)
* iii) Exocrine pancreatic insufficiency, defined as pancreatic steatorrhea markedly reduced by enzyme supplementation
* iv) Histological verification of CP
* A probable diagnosis of CP is established by one or more of the following additional criteria:
* i) Mild ductal alterations (according to the Cambridge classification)
* ii) Recurrent or persistent pseudocysts
* iii) Pathological test of pancreatic exocrine function (such as faecal elastase-1 test, secretin test, secretin-pancreozymin test)
* iv) Diabetes mellitus
* Abdominal pain of presumed pancreatic origin (i.e., upper abdominal pain radiating to the back).
* Evidence of ongoing pancreatic inflammatory activity, with an inflammatory pancreatic flare occurring one or more times within the past six months. An inflammatory pancreatic flare is defined as an exacerbation of pancreatic pain in combination with one or more of the following criteria:
* i) Plasma amylase levels elevated 2-fold or more than the participant's usual amylase level.
* ii) Elevated plasma levels of CRP 2-fold the upper normal level without suspicion of other sources such as infection.
* iii) Signs of pancreatic inflammation on cross-sectional imaging.
* ≥ 18 years of age
* The participant must be able to read and understand the informed consent forms.
* The participant is willing and able to comply with the scheduled visits, treatment plan, and other trial procedures.

Exclusion Criteria:

* End-stage CP indicated by severe pancreatic atrophy defined as segmented pancreas volume <20 ml on the latest available cross-sectional imaging examination (Computed Tomography (CT) or MRI).
* Pancreatic duct obstruction by a stricture and/or stone amendable to endoscopic or surgical treatment. Patients with previous pancreatic duct decompression procedures are allowed to participate.
* Ongoing alcohol or substance abuse. The patient must document abstinence from alcohol and substance abuse for the preceding six months prior to study enrolment. Recreational alcohol consumption within the safety limits recommended by the National Danish Health Authorities (i.e., max. ten units of alcohol per week) is allowed.
* Active or recurrent infections.
* Untreated ulcers in the gastrointestinal tract (however, those who have undergone proper treatment and one month has elapsed with no recurrence of symptoms will not be excluded).
* Known hypersensitivity to Tocilizumab.
* Positive test for Tuberculosis during screening
* Positive test for Hepatitis during screening
* Severe liver disease, indicated by ALT with >5 upper normal limits.
* Thrombocytopenia (platelet count < 50 x 109/L).
* Neutropenia (neutrophil count <2 x 109/L).
* Pregnancy and no contraception use, fertile women (<55 years) must provide a urine sample for pregnancy test upon inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
The Comprehensive Pain Assessment Tool Short Form (COMPAT-SF) Questionnaire | The intervention period is 24 weeks (assessed every 4 weeks from baseline to finalization)
  The between-group difference (tocilizumab vs. placebo) of the change from baseline in the COMPAT-SF score at 24 weeks. The COMPAT-SF score is noramlized on a 0-100 score. Higher scores indicate a higher degree of pain.

SECONDARY OUTCOMES:
Global Quality of Life Score (EORTC-QLQ-C30) | The intervention period is 24 weeks (assessed at weeks 0, 12, and 24)
  The between-group difference in the Global Quality of Life Score from baseline in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C-30 (EORTC-QLQ-C30) questionnaire at 24 weeks. The global quality of life score range from 0 to 100. A high score on the Global Quality of Life score represents a high level of life quality.
Physical Functional Score (EORTC-QLQ-C30) | The intervention period is 24 weeks (assessed at weeks 0, 12, and 24)
  The between-group difference in Physical Functional Score from baseline in the EORTC-QLQ-C30 questionnaire at 24 weeks. The physical functional score ranges from 0 to 100. A high score on the functional scales represents a high level of daily functioning.
Role Functional Score (EORTC-QLQ-C30) | The intervention period is 24 weeks (assessed at weeks 0, 12, and 24)
  The between-group difference in Role Functional Score from baseline in the EORTC-QLQ-C30 questionnaire at 24 weeks. The role functional score ranges from 0 to 100 A high score on the functional scales represents a high level of daily functioning.
Cognitive Functional Score (EORTC-QLQ-C30) | The intervention period is 24 weeks (assessed at weeks 0, 12, and 24)
  The between-group difference in Cognitive Functional Score from baseline in the EORTC-QLQ-C30 questionnaire at 24 weeks. The cognitive functional score ranges from 0 to 100. A high score on the functional scales represents a high level of daily functioning.
Emotional Functional Score (EORTC-QLQ-C30) | The intervention period is 24 weeks (assessed at weeks 0, 12, and 24)
  The between-group difference in Emotional Functional Score from baseline in the EORTC-QLQ-C30 questionnaire at 24 weeks. The emotional functional score ranges from 0 to 100. A high score on the functional scales represents a high level of daily functioning.
Social Functional Score (EORTC-QLQ-C30) | The intervention period is 24 weeks (assessed at weeks 0, 12, and 24)
  The between-group difference in Social Functional Score from baseline in the EORTC-QLQ-C30 questionnaire at 24 weeks. The social functional score ranges from 0 to 100. A high score on the functional scales represents a high level of daily functioning.
Symptom Burden Score (EORTC-QLQ-C30) | The intervention period is 24 weeks (assessed at weeks 0, 12, and 24)
  The between-group difference in Symptom Score from baseline in the EORTC-QLQ-C30 questionnaire at 24 weeks. The symptom burden score ranges from 0 to 100. A high score for the symptom items represents a high level of symptomatology.
Pain severity Score (modified BPI) | The intervention period is 24 weeks (assessed at weeks 0, 12, and 24)
  The between-group difference in Pain severity score from baseline in the modified Brief Pain Inventory at 24 weeks. The pain severity score is rated on a visual analogue scale (VAS), 0 = no pain, 10 = worst pain imaginable), based on four pain severity items. Higher scores reflect more severe pain.
Pain Interference Score (modified BPI) | The intervention period is 24 weeks (assessed at weeks 0, 12, and 24)
  The between-group difference in Pain Interference score from baseline in the modified Brief Pain Inventory at 24 weeks. The pain interference score is rated on a VAS, 0 = no pain, 10 = worst pain imaginable, based on seven pain interference items. Higher scores reflect more pain interference with daily life.
Average Daily Pain Score (modified BPI) | The intervention period is 24 weeks (assessed at weeks 0, 12, and 24)
  The between-group difference in Average Daily Pain score from baseline in the modified Brief Pain Inventory at 24 weeks. The average daily pain score ranges is rated on a VAS-scale, 0-10, 0 = no pain, and 10 = worst pain imaginable.
Patient's Global Impression of Change (PGIC) Questionnaire | The intervention period is 24 weeks (assessed at week 24)
  The between-group difference in the PGIC questionnaire, a self-reporting seven-point rating scale (points from 1-7) on how the participant experiences treatment change from baseline at 24 weeks. Higher score corresponds to improvement.
CP Prognosis Score | The intervention period is 24 weeks (assessed at weeks 0 and 24)
  The between-group difference in the CP prognosis score from baseline at 24 weeks. The CP prognosis score ranges from 5-15 points. Higher scores indicates higher risk of readmission to hospital.
Number of patient using prescription opioids for pain control | The intervention period is 24 weeks (continuously throughout the entire study)
  Opioid use (yes, no, binary answer) continuously through the entire study
Daily opioid dose for patients using prescription opiods | The intervention period is 24 weeks (continuously throughout the entire study)
  The between and within-group difference of opioid dose (continuous variable in mg of moprhine equivalent) in patients, from baseline at 24 weeks.
Number of patient using weak analgesics for pain control | The intervention period is 24 weeks (continuously throughout the entire study)
  Weak analgesic use (yes, no, binary answer) continuously through the entire study
Daily weak analgesics dose for patients | The intervention period is 24 weeks (continuously throughout the entire study)
  The between and within-group difference of weak analgesic dose (continuous variable in mg) in patients, from baseline at 24 weeks.
Frequency of adverse events (Patient Diary) | The intervention period is 24 weeks (continuously throughout the entire study)
  The frequency of adverse events from baseline at 24 weeks.

OTHER OUTCOMES:
Levels of soluble inflammation biomarker | The intervention period is 24 weeks (samples drawn at weeks 0, 4, 8, 16, and 24)
  The investigators plan to use an O-link multiplex platform to examine changes in soluble inflammatory biomarker levels, including several cytokines and chemokines.
Levels of soluble fibrosis biomarker | The intervention period is 24 weeks (samples drawn at weeks 0, 4, 8, 16, and 24)
  The investigators plan to use an O-link multiplex platform to examine changes in soluble fibrosis biomarker levels, from baseline at 24 weeks.
Levels of soluble Biomarker of Macrophage Activation | The intervention period is 24 weeks (samples drawn at weeks 0, 4, 8, 16, and 24)
  Macrophage activation biomarkers will be analyzed using enzyme-linked immunosorbent assays (ELISAs) levels, from baseline at 24 weeks.
Levels of key Inflammatory Mediator | The intervention period is 24 weeks (samples drawn at weeks 0, 4, 8, 16, and 24)
  For the key inflammatory mediator, found in above mentioned analysis, the investigators will confirm the analyses using ELISAs levels from baseline at 24 weeks.
Pancreatic inflammation (imaging) | The intervention period is 24 weeks (conducted at weeks 0 and 24)
  The between and within-group difference of diffusion-weighted imaging for inflammation using multiparametric pancreatic MRI at baseline and after 24 weeks.
Pancreatic fibrosis (imaging) | The intervention period is 24 weeks (conducted at weeks 0 and 24)
  The between and within-group difference of fibrosis detection using T1 mapping multiparametric pancreatic MRI parameters at baseline and after 24 weeks.
Pancreatic morphology (imaging) | The intervention period is 24 weeks (conducted at weeks 0 and 24)
  The between and within-group difference of conventional anatomic imaging using multiparametric pancreatic MRI at baseline and after 24 weeks.
Pancreatic duct morphology (imaging) | The intervention period is 24 weeks (conducted at weeks 0 and 24)
  The between and within-group difference of pancreatic duct morphology using Magnetic resonance cholangiopancreatography (MRCP) at baseline and after 24 weeks.
Biliary duct morphology (imaging) | The intervention period is 24 weeks (conducted at weeks 0 and 24)
  The between and within-group difference of biliary duct morphology using MRCP at baseline and after 24 weeks.
P-QST: PinPrick (Temporal summation) | The intervention period is 24 weeks (performed at weeks 0 and 24)
  The pancreatic quantitative sensory testing (P-QST) is used to characterize pain processing and comprises different experimental pain stimuli:
  PinPrick test: A pinprick stimulator 256 mN (MRC Systems GmbH, Germany) will be used to perform the pinprick test. The patient is asked to rate the pain sensitisation using the VAS score after a single pinprick stimulus and after ten repetitive stimuli (applied with an interstimulus interval of 1 second). Two test areas are assessed: the dominant forearm and the anterior TH10 dermatome. The score is reported on a VAS score from 0 to 10. Higher scores indicate higher pain tolerance.
P-QST: Pain Pressure thresholds | The intervention period is 24 weeks (performed at weeks 0 and 24)
  The P-QST is used to characterize pain processing and comprises different experimental pain stimuli:
  Pain pressure test: Pressure algometry is performed with a handheld pressure algometer (Type2, Somedic production AB, Sweden) and performed in four dermatomes and five locations: C5 (the clavicle), TH10 (the back and abdomen), L1 (the anterior superior iliac spine), and L4 (straight thigh). The probe has a surface area of 1cm2. Pressure will be increased at a rate of 30 kPa/sec until prespecified thresholds (i.e., pain detection threshold (PDT) and pain tolerance threshold (PTT)) are reached. The assessment parameters are the imposed pressure (kPa) at the PDT and PTT.
P-QST: Cold Pressor | The intervention period is 24 weeks (performed at weeks 0 and 24)
  The P-QST is used to characterize pain processing and comprises different experimental pain stimuli:
  Cold pressor test: The patient's hand is immersed in cold water (approximately two degrees Celsius) for 120 seconds. At 40, 80, and 120 seconds, the patient is asked to rate the pain sensation using a VAS score. If the patient cannot keep their hand in the water for 120 seconds, the duration is noted, and the VAS score at the time they withdraw their hand is used as the maximum score. The assessment parameters are the cold pressor endurance time (seconds) and the evoked pain responses on a visual analog scale (VAS) score, 0 = no pain and 10 = worst pain imaginable. Lower values indicate higher pain tolerance.
P-QST: Conditioned Pain Threshold | The intervention period is 24 weeks (performed at weeks 0 and 24)
  The P-QST is used to characterize pain processing and comprises different experimental pain stimuli:
  Conditioned pain modulation test is conducted using a pain pressure algometer, and the PTT is assessed at 15 cm above the patella in the L4 dermatome on the nondominant side before and after the cold pressor test is performed.
  The imposed pain pressure tolerance threshold is reported as kPa, with a minimum of 0, and no upper limit. Higher scores indicate higher pain tolerance.
Electroencephalography (EEG) analysis | The intervention period is 24 weeks (assessed at weeks 0 and 24)
  While performing the P-QST, the investigators measure EEG and ECG before and after the cold pressor test.
  A standard EEG electrode Cap Kit (EEG Electrode Cap Kit - OpenBCI Online Store) with ten electrodes is employed for these measurements.The Texas Instrument ADS1299 biopotential measurements system will be used for EEG and ECG recordings. This system is already being used in mobile brain-computer interfaces, and its signals are comparable to those of standard systems that can work in hospital settings. The EEG signals are transmitted wirelessly to an Android mobile telephone and stored for further processing.
  The results will be used to model connectivity between brain centres as well as the dominating centres of the brain. EEG power will be assessed in the Delta, Theta, Alpha, Beta, and Gamma bands between 1 and 70 Hertz. Finally, inverse modelling will be conducted to explore the dominating centres of brain activity.
Electrocardiographic (ECG) frequency domain | The intervention period is 24 weeks (assessed at weeks 0 and 24)
  Four conventional ECG electrodes (Neurolink 700) is employed for these measurements. The ECG signals are transmitted wirelessly to an Android mobile telephone and stored for further processing.
  Frequency domains of heart variablity will be assessed using ECG,this involve Fast Fourier transformation of the Blackman Harris window included very low frequency (VLF), low frequency (LF), high frequency (HF), total power (TP), and the ratios LF/HF.
ECG time domain | The intervention period is 24 weeks (assessed at weeks 0 and 24)
  Four conventional ECG electrodes (Neurolink 700) is employed for these measurements. The ECG signals are transmitted wirelessly to an Android mobile telephone and stored for further processing.
  Time domains of heart variablity will be assessed using ECG, this involve determining the mean RR interval, standard deviation of RR interval, heartbeat rate (HR), and root mean squared difference of successive normal RR intervals (RMSSD).

CONTACTS AND LOCATIONS:
Overall Officials: Søren S Olesen, MD, Ph.D., Principal Investigator — Mech-Sense, Department of Gastroenterology, Aalborg University Hospital
Locations (1):
- Centre for Pancreatic Diseases and Mech-Sense research laboratory, Aalborg University Hospital, Aalborg, North Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No
Access to the data is available upon reasonable request.